CLINICAL TRIAL: NCT06508788
Title: Combinación Del láser Vaginal Con un Gel Niosomal Hidratante y Reparador en el Tratamiento Del síndrome Genitourinario en Pacientes oncológicas
Brief Title: Combination of the Vaginal Laser With a Moisturizing and Repairing Niosomal Gel in the Treatment of Genitourinary Syndrome in Oncology Patients
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Carlos Ortega-Expósito, Principal Investigator, Hospital Universitari de Bellvitge
Other Study IDs: ICPS010/24
Record Dates: First submitted 2024-07-15; First posted 2024-07-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: Genitourinary Syndrome of Menopause; CO2 laser
MeSH Terms: interventions — Lasers, Gas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CO2 laser cohort: Patients with a history of oncology and for whom a diagnosis of genitourinary syndrome is established and who are not eligible for treatment with hormonal therapy
  Interventions: Device: CO2 laser

INTERVENTIONS:
Device: CO2 laser — Application of CO2 vulvo-vaginal laser according to standard therapy and moisturizing gels

SUMMARY:
Vaginal laser together with the use of moisturizing and repairing gels could be an effective therapy for the treatment of genitourinary syndrome in women with a history of neoplasia in whom the use of estrogens is not recommended.

The purpose of this study is to evaluate the effectiveness of vaginal laser together with adjuvant treatment with a hydrating and repairing niosomal gel as a beneficial treatment in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established SGM diagnosis.
* Patients with a history of neoplasia in whom the use of estrogens as the first alternative for the treatment of GMS is not recommended.

Exclusion Criteria:

* Patients with concomitant vulvovaginal pathology.
* Patients with a diagnosis of pelvic organ prolapse grade II or greater.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an established SGM diagnosis who have a history of neoplasia in whom the use of estrogens as the first alternative for the treatment of GMS is not recommended.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 12 months
  To evaluate the effectiveness of CO2 vaginal laser together with adjuvant treatment with a hydrating and repairing niosomal gel as a beneficial treatment in patients with a history of neoplasia in whom the use of estrogens is not recommended

SECONDARY OUTCOMES:
Security | 12 months
  To determine the safety (side effects) of vaginal laser therapy
Duration | 12 months
  To determine the durability of the effects produced by vaginal laser therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos, L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No